CLINICAL TRIAL: NCT02824029
Title: A Phase II Multicenter Single Arm Study to Evaluate the Efficacy and Safety of Single Agent Bruton's Tyrosine Kinase Inhibitor, Ibrutinib, in Patients With Relapsed Refractory Classical Hodgkin's Lymphoma
Brief Title: Ibrutinib in Treating Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dipenkumar Modi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-033; NCI-2016-00879 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-033 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2016-06-20; First posted 2016-07-06 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Classical Hodgkin Lymphoma; Recurrent Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ibrutinib) (Experimental): Patients receive ibrutinib PO QD. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial evaluates how effective 560 mg of ibrutinib taken by mouth daily is in the treatment of classical Hodgkin lymphoma which recurs or does not respond to initial treatment. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth, by altering the environment around the tumor or by affecting the immune system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the antitumor efficacy of single agent ibrutinib as measured by the overall response rate in patients with relapsed/refractory Hodgkin's lymphoma who have relapsed or not responded to chemotherapy, immunotherapy and/or radiation.

SECONDARY OBJECTIVES:

I. To assess duration of tumor control including duration of response (DOR) II. To assess progression free survival (PFS). III. To assess the safety and tolerability of 560mg of ibrutinib in Hodgkin lymphoma (HL) patients.

TERTIARY OBJECTIVES:

I. To assess the mechanism(s) by which ibrutinib may be active in patients with classical Hodgkin lymphoma (cHL) by the correlation of potential biomarkers with clinical outcomes.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days then every 9 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria

* Patients with relapsed or refractory classical HL who have previously received autologous stem cell transplant and/or allogeneic stem cell transplant. Patients must have received prior autologous stem cell transplant at least 12 weeks (3 months) before the first dose of ibrutinib and/or allogeneic stem cell transplant must have been completed at least 6 months prior to the first dose of Ibrutinib. OR
* Patients with relapsed or refractory HL who have failed at least 2 lines of prior therapy and are not eligible for autologous stem cell transplant due to:

  * Inability to achieve a CR or PR prior to transplant
  * Age or comorbid conditions
  * Inability to collect stem cells
* Completion of any prior treatment with radiation, chemotherapy, biologics, and/or other investigational agents at least 4 weeks prior to the first dose of ibrutinib. Patients must have completed any prior immunotherapy (e.g., rituximab or PD-1 inhibition) or antibody drug conjugate therapy (e.g. brentuximab vedotin) at least 4 weeks prior to the first dose of ibrutinib in the absence of clear disease progression.
* Prior treatment with at least 2 lines of therapy for HL including brentuximab vedotin. In those patients who cannot receive brentuximab vedotin, treatment with 2 prior therapeutic regimens is sufficient.
* Fluorodeoxyglucose (FDG)-avid disease by PET and measurable disease of at least 1.5 cm in minimum dimension by CT scan with contrast, as assessed by the site radiologist.
* Adequate hematologic function independent of transfusion and growth factor support for at least 7 days prior to screening and randomization, with the exception of PEGylated GCSF (pegfilgrastim) and darbopoeitin which require at least 14 days prior to screening and randomization defined as:

  * Absolute neutrophil count >750 cells/mm3 (0.75 x 109/L).
  * Platelet count >50,000 cells/mm3 (50 x 109/L).
  * Hemoglobin >8.0 g/dL.
* Adequate hepatic and renal function defined as:

  * Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN).
  * Estimated Creatinine Clearance ≥30 ml/min (Cockcroft-Gault)
  * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
* PT/INR <1.5 x ULN and PTT (aPTT) <1.5 x ULN.
* Men and women ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Female subjects who are of non-reproductive potential (i.e., post-menopausal by history-no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female subjects of childbearing potential must have a negative serum pregnancy test upon study entry.
* Male and female subjects who agree to use highly effective methods of birth control (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) during the period of therapy and for 90 days after the last dose of study drug
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Prior allogeneic Stem cell transplant within 6 months.
* Active GVHD or concurrent treatment with immunosuppressive medications as prophylaxis for GVHD
* Previous therapy with BTK inhibition
* Known cerebral/meningeal disease
* Nodular lymphocyte predominant Hodgkin's Lymphoma subtype
* Concurrent therapy with other systemic anti-neoplastic or investigational agents
* Patients with a known hypersensitivity to any excipient contained in the drug formulation
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for

    ≥3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine A, tacrolimus, etc., or chronic administration [>14 days] of >20 mg/day of prednisone) within 28 days of the first dose of study drug.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Recent infection requiring systemic treatment that was completed ≤14 days before the first dose of study drug.
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4), grade ≤1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV). Subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* Any uncontrolled active systemic infection
* Major surgery within 4 weeks of first dose of study drug.
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Concomitant use of warfarin or other Vitamin K antagonists.
* Requires treatment with a strong cytochrome P450 (CYP) 3A4/5 inhibitor
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification
* Lactating or pregnant
* Unwilling or unable to participate in all required study evaluations and procedures.
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Potential subjects must be willing and able to adhere to the following prohibitions and restrictions during the course of the study to be eligible for participation. During the study, subjects should avoid consuming food and beverages containing grapefruit or Seville oranges as these contain certain ingredients that inhibit CYP3A4/5 enzymes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-06; Primary Completion 2023-05-12 (Actual); Study Completion 2025-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dipenkumar Modi, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (4):
- United States (4):
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - University of Tennessee, Knoxville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Muqbil I, Chaker M, Aboukameel A, Mohammad RM, Azmi AS, Ramchandren R. Pre-clinical anti-tumor activity of Bruton's Tyrosine Kinase inhibitor in Hodgkin's Lymphoma cellular and subcutaneous tumor model. Heliyon. 2019 Aug 31;5(8):e02290. doi: 10.1016/j.heliyon.2019.e02290. eCollection 2019 Aug. PMID 31508518

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ibrutinib)
Started | 28
Completed | 0
Not Completed | 28
Not completed — Didn't receive treatment | 2
Not completed — Patient decision to discontinue treatment | 3
Not completed — Non-compliant | 5
Not completed — Progression of disease | 15
Not completed — Inadequate response to therapy | 2
Not completed — Possible progression per treating physician | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 37.5 [23 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 20
  Race: Black or African American | 3
  Race: Other | 1
  Race: Unknown or Not reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 28
Stage at Enrollment [Count of Participants; unit: Participants] — Using Ann Arbor Staging System. The higher the stage number, the more the lymphoma has spread.
  Participants
    II | 4
    III | 11
    IV | 8
    Unknown | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) defined as the proportion of participants having a complete (CR) and partial (PR) response. A one-sample binomial test will be used to assess ORR.
Time Frame: From date of study entry to date of progression or death up to 24 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 21
Proportion of participants | 0.05 [0.002 to 0.23]

2. Secondary Outcome: Duration of Response (DOR)
Description: Kaplan-Meier estimate of median DOR will be reported with 95% confidence intervals.
Time Frame: From date of documented tumor response, CR or PR, to date of disease progression or death, up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 1
months | 5.6 [NA to NA] — Since only one patient achieved PR, none achieved CR, the confidence interval is not evaluable.

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Kaplan-Meier estimate of median PFS will be reported with 95% confidence intervals.
Time Frame: From date of study entry to date of progression or death up to 24 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 21
months | 4.6 [1.9 to 6.4]

ADVERSE EVENTS:
Time Frame: From date of study entry to date of progression or death up to 27 months
Arm/Group | Treatment (Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 8/26
Serious Adverse Events (participants affected / at risk) | 5/26
Other Adverse Events (participants affected / at risk) | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=26)
Dental: teeth (Gastrointestinal disorders) | 1 (1)
Obstruction, GI (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=26)
Edema (Blood and lymphatic system disorders) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 4 (6)
Palpitations (Cardiac disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 11 (12)
Gastrointestinal (Gastrointestinal disorders) | 2 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 5 (5)
Mucositis/stomatitis (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 11 (20)
Pain - Abdomen NOS (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)
Xerostomia (Gastrointestinal disorders) | 3 (3)
Constitutional Symptoms (General disorders) | 2 (2)
Fatigue (General disorders) | 7 (8)
Fever (General disorders) | 3 (4)
Insomnia (General disorders) | 4 (4)
Pain (General disorders) | 6 (7)
Syndromes (General disorders) | 2 (2)
Allergic rhinitis (Immune system disorders) | 3 (3)
Infection (Infections and infestations) | 5 (5)
Hemorrhage (Injury, poisoning and procedural complications) | 2 (2)
ALT, SGPT (Metabolism and nutrition disorders) | 4 (4)
AST, SGOT (Metabolism and nutrition disorders) | 4 (4)
Creatinine (Metabolism and nutrition disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain - Back (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 7 (9)
Pain - Neck (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 4 (7)
Mood alteration - Anxiety (Nervous system disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 5 (5)
Pain - Head/headache (Nervous system disorders) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary/respiratory (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 4 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT02824029/Prot_SAP_000.pdf